CLINICAL TRIAL: NCT04843241
Title: Test of Reliability and Validation of Neck Disability Index Questionnaire in Local Languages of Pakistan
Brief Title: Translation of Neck Disability Index Into Local Pakistani Languages of Pakistan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/00934 Syed Hashir Ali
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Neck Pain
Keywords: Neck Pain; Neck Disability Index; Tool Translation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to translate the neck disability index (NDI) questionnaire into Pushto, Punjabi, Sindhi and Balochi versions and o test the validity & reliability of translated versions of NDI among neck pain patients in Pakistan.

DETAILED DESCRIPTION:
The Neck Disability Index is a state-unambiguous instrument for the description of a disability. It is revised from the Oswestry Low Back Pain Questionnaire It contains 10 items mentioning various activities (personal care, lifting, driving, work, sleeping, concentration, reading, recreation) and pain (pain intensity, headache) with 6 conceivable answers for each item. Patients are educated to choose only one answer which most closely suits their condition at the current time. The score of each item ranges between 0 (no pain and no functional limitation) and 5 (worst pain and maximal limitation) that lead to the total score of 0 (no disability) to 50 (totally disabled), as 0-4 points (no disability), 5-14 points (10-28% disability), 15-24 points (30-48% disability), 25-34 points (50-64% disability) and 35-50 points (70-100% disability). The meantime to fill the questionnaire is 3-7.8 minutes. The NDI showed high validity and reliability for patients with neck pain.

By this study, the accuracy and reproducibility of the translated versions of NDI questionnaires will be enhanced and thus can create a useful measure to obtain data from culturally/linguistically diverse people belonging to different ethnic background as in Pakistan. It will create trustworthiness among clinicians and researchers to utilize the tool as a measure of what it is supposed to measure.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical neck pain
* Participants belonging to Urdu, Pushto, Punjabi, Sindhi and Balochi speaking class
* Participants from inpatient and outpatient department of hospitals
* participants should complete the questionnaire in their respective language without the help

Exclusion Criteria:

* Healthy Individuals
* Pathological neck pain
* Traumatic cervical or neck injuries
* Participants with disability due to any structural/ congenital cause

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To meet inclusion criteria participants diagnosed with neck pain, clinically stable, and able to read the local language version of NDI. Then patient response will be checked on the translated version
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Translation of the Neck Disability Index questionnaire into Pushto, Punjabi, Sindhi and Balochi versions | 6 months
  The Neck Disability Index is a state-unambiguous instrument for the description of a disability. It is revised from the Oswestry Low Back Pain Questionnaire It contains 10 items mentioning various activities (personal care, lifting, driving, work, sleeping, concentration, reading, recreation) and pain (pain intensity, headache) with 6 conceivable answers for each item, so translation for this NDI is to be done into regional languages of Pakistan through a rigorous and approved process. The minimum and maximum possible scores could be 0 and 50. The higher the score more the disability is there.

SECONDARY OUTCOMES:
Test the validity & reliability of translated versions of Neck Disability Index among neck pain patients in Pakistan | 6 months
  To determine reliability and validity of cross-culturally adapted and the translated NDI versions in patients with neck pain of respective languages۔ Reliability or reproducibility refers to the ability of a measure to produce the same results when administered at two or more interval between different visits of the patient and validity is how accurate the results are. Thus these both are to measured through various parameters to validate the translated versions as appropriate and applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Margalla Rehabilitation Center, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rathore FA, Attique R, Asmaa Y. Prevalence and Perceptions of Musculoskeletal Disorders Among Hospital Nurses in Pakistan: A Cross-sectional Survey. Cureus. 2017 Jan 26;9(1):e1001. doi: 10.7759/cureus.1001. PMID 28280654
- [Background] Andersson HI, Ejlertsson G, Leden I, Rosenberg C. Chronic pain in a geographically defined general population: studies of differences in age, gender, social class, and pain localization. Clin J Pain. 1993 Sep;9(3):174-82. doi: 10.1097/00002508-199309000-00004. PMID 8219517
- [Background] Howell ER. The association between neck pain, the Neck Disability Index and cervical ranges of motion: a narrative review. J Can Chiropr Assoc. 2011 Sep;55(3):211-21. PMID 21886283
- [Background] Farooq MN, Mohseni-Bandpei MA, Gilani SA, Hafeez A. Urdu version of the neck disability index: a reliability and validity study. BMC Musculoskelet Disord. 2017 Apr 8;18(1):149. doi: 10.1186/s12891-017-1469-5. PMID 28388888